CLINICAL TRIAL: NCT03212456
Title: Evaluation of Post-operative Biochemical Recurrence in Patients Submitted to Radical Prostatectomy Under General Opioid-free Anesthesia Compared to Conventional General Anesthesia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Instituto do Cancer do Estado de São Paulo (Other)
Responsible Party: Principal Investigator, Felipe Rangel, MD, Anesthesiologist, principal investigator, Instituto do Cancer do Estado de São Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NP 834/15
Record Dates: First submitted 2017-04-10; First posted 2017-07-11 (Actual); Last update posted 2020-07-29 (Actual); Status verified 2020-07

CONDITIONS: Prostate Cancer
Keywords: general anesthesia; cancer recurrence; opioids analgesics; neoplasm
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasms | interventions — Ropivacaine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Opioid-free (Experimental): The patients of this group will receive opioid-free anesthesia
  Interventions: Drug: opioid-free group; Procedure: transversus abdominal plane block with ropivacaine
- Non opioid-free (Active Comparator): The patients in this group will receive the same induction and maintenance drugs of the experimental group but with fentanyl 3 - 5 mcg/kg on induction and during the procedure as needed.
  Interventions: Drug: Opioid Group; Procedure: transversus abdominal plane block with placebo

INTERVENTIONS:
Drug: opioid-free group — We'll study if the opioid-free anesthesia can reduce the biochemical recurrence of prostate cancer.
  Arms: Opioid-free
Drug: Opioid Group — This group will receive fentanyl in the induction of anesthesia.
  Arms: Non opioid-free
Procedure: transversus abdominal plane block with ropivacaine — The opioid-free group will receive transversus abdominal plane block with ropivacaine 0,375% 20 ml each side
  Arms: Opioid-free
Procedure: transversus abdominal plane block with placebo — the non-opioid free group will receive transversus abdominal plane block with physiological solution 0,9% 20 ml each side
  Arms: Non opioid-free

SUMMARY:
The use of opioids facilitates angiogenesis and has a proven action in the immune system, mainly in the reduction of natural killer cell activity, favoring the migration of neoplastic cells and inhibiting humoral and cellular immunity. These factors may contribute to recurrence and tumor metastasis.

Therefore, could opioid-free anesthesia help reduce tumor recurrence? This is a prospective randomized controlled clinical trial in which patients undergoing radical prostatectomy will be evaluated by conventional means, which have moderate and high D'Amico criteria for tumor recurrence.

In the operating room, patients will be monitored, receive peripheral venoclysis and then randomized into two groups: in group I, the anesthetic induction will be done with pre oxygenation with 100% O2, propofol, cisatracurium, lidocaine and fentanyl; In group II the induction will be done with the same doses of propofol, cisatracurium, lidocaine and placebo.

In both groups maintenance of general anesthesia will be with propofol 1% target infusion controlled with model of Marsh target-controlled infusion plasma between 2.0 and 3.0 mcg / ml, ketamine, lidocaine and dexmedetomidine.

Both groups will receive blockade of the transverse plane of the ultrasound guided ultrasound, group I with placebo (saline 0.9% 20 ml on each side) and group II with ropivacaine 0.375% 20 ml on each side. And the postoperative analgesia will be based on anti-inflammatory and opioid analgesics (pca of morphine) according to the analgesic pain scale of the patients.

In the postoperative period, patients will be followed up for 2 years with serial doses of prostate specific antigen (PSA) to diagnose tumor recurrence (2 PSA measures> 0.2 ng / ml) and will be evaluated in relation to analgesia, need for analgesia of Rescue with morphine, satisfaction with the anesthetic technique, adverse effects (nausea and vomiting).

The primary objective is to evaluate tumor biochemical recurrence after radical prostatectomy in patients undergoing opioid anesthesia compared to patients anesthetized without opioids. The secondary objectives are to evaluate the quality of analgesia with the two techniques, patient satisfaction with perioperative period, quality of anesthetic recovery and adverse effects (nausea and vomiting, pruritus and drowsiness).

Thus, to answer the hypothesis raised, 146 patients will be needed (73 in each group).

ELIGIBILITY:
Inclusion Criteria:

* Prostate Cancer;
* Intermediate to high risk of recurrence by D'Amico criteria (Gleason scale > or = 7; PSA > or = 10)

Exclusion Criteria:

* Patient refuse;
* atrioventricular blockade;
* Coagulopathy;
* Other procedure at same time.

Ages: 40 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2017-01-12 (Actual); Primary Completion 2020-09-30 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
Biochemical recurrence of prostate cancer | Up to 2 years after the date of the surgery
  It's going to be measured the prostate specific antigen in 4 times after the date of the surgery( 6 months, 1 year, 1 and a half year and 2 years after the surgery) to compare elevations between the two groups.

SECONDARY OUTCOMES:
Neutrophil-to-lymphocyte ratio | 24 hour postoperatively
  Compare the peutrophil-to-lymphocyte ratio preoperatively and with 24 hour postoperatively between the two groups to study about inflammation.
visual analogue pain score in the post-anaesthesia care unit | Up to 2 hours postoperatively
  Compare the pain scale between the two groups in the delivery of post-anaesthesia care unit
Rescue Morphine | Up to 2 hours postoperatively
  compare the total dosis needed for pain at delivery post-anaesthesia care unit
Satisfaction with anesthesia technique | Up to 2 hours postoperatively
  compare the satisfaction (a scale from 01 to 10) with anesthesia technique between the two groups at delivery of post-anaesthesia care unit
adverse outcomes | Up to 2 hours postoperatively
  compare the postoperative adverse outcomes (such as nausea, pruritus, somnolence) between the two groups at delivery of post-anaesthesia care unit

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto do Cancer do Estado de Sao Paulo - Icesp, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
The following data will be available: which group the patient were randomized; BMI; PSA preoperatively, 6 months, 1 year, 1,5 year and 2 years; prostate volume; gleason scale; neutrophil-to-lymphocyte ratio preoperatively and postoperatively; bleeding; intraoperative hydration; amount of opioids in the intraoperative period; VAS pain scale in the PACU and morphine dosis in the PACU

REFERENCES:
- [Derived] Rangel FP, Auler JOC Jr, Carmona MJC, Cordeiro MD, Nahas WC, Coelho RF, Simoes CM. Opioids and premature biochemical recurrence of prostate cancer: a randomised prospective clinical trial. Br J Anaesth. 2021 May;126(5):931-939. doi: 10.1016/j.bja.2021.01.031. Epub 2021 Mar 10. PMID 33712224